CLINICAL TRIAL: NCT06025513
Title: A Phase 1 Study to Assess the Safety and Efficacy of Embrace, De-tensioning Patch, in Subjects With Type 1 Diabetes and Lipohypertrophy (LH)
Brief Title: De-tensioning Patch, in Subjects With Type 1 Diabetes and Lipohypertrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neodyne Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA006
Record Dates: First submitted 2023-08-23; First posted 2023-09-06 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Insulin Resistance; Lipohypertrophy
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Pre / Post comparison with device treatment for 16 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- embrace patch treatment (Experimental): Insulin PK/PD before and after treatment with embrace patch
  Interventions: Device: Embrace Patch

INTERVENTIONS:
Device: Embrace Patch — Tension offloading skin patch

SUMMARY:
This is a single-center, single-cohort, open, repeated-application study. Baseline assessments will include a Hyperinsulinemic clamp after injection of 0.15 U/kg body weight of insulin lispro in the target LH lesion, as well as a Mixed Meal Tolerance Test (MMTT) with pre-meal insulin injected into the LH lesion. Subjects will discontinue their basal insulin for 2-3 days after the Continuous glucose monitor (CGM) study ends, prior to admission to the research center ("wash-out"). After release from the research center, subjects will wear the Embrace over the target LH lesion for 16 weeks. At the beginning of week 17, the clamp and MMTT will be repeated, after which participants will again wear an unblinded CGM for ~6 days with injections only in the target LH lesion when applying an Embrace patch with a hole. A needle biopsy will be taken from the LH lesion at baseline and again at study completion.

DETAILED DESCRIPTION:
This is a single-center, single-cohort, open, repeated-application study. Baseline assessments will include a Hyperinsulinemic clamp after injection of 0.15 U/kg body weight of insulin lispro in the target LH lesion, as well as a Mixed Meal Tolerance Test (MMTT) with pre-meal insulin injected into the LH lesion. However, before admission to the research center, unblinded CGM is worn for ~13 days (day 1 is discarded to avoid variability, day 2-7 bolus injections in Normal Tissue (NAT) and day 8-13 bolus injections in target LH) as outpatients. Subjects will discontinue their basal insulin for 2-3 days after the CGM study ends, prior to admission to the research center ("wash-out"). After release from the research center, subjects will wear the Embrace over the target LH lesion for 16 weeks, reapplying the patch every week and avoiding any injections in the target LH lesion. Basal insulin is injected only in NAT away from the LH site. At the beginning of week 17, the clamp and MMTT will be repeated, after which participants will again wear an unblinded CGM for ~6 days (again, day 1 is discarded) with injections only in the target LH lesion when applying an Embrace patch with a hole. A needle biopsy will be taken from the LH lesion at baseline and again at study completion.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent obtained before any trial-related activities. Trial-related activities are any procedures that would not have been done during normal management of the subject.
2. Subject with type 1 diabetes for at least 3 years
3. One or more palpable lipohypertrophy lesions in the abdominal area, the largest of which has a minimum size of 3.0 cm and a maximum size of 12.0 cm (longest axis) as confirmed by ultrasound.
4. Treated with multiple daily injections (≥3) of insulin for at least 2 years or continuous subcutaneous insulin infusion for at least 1 year.
5. Subject is willing and able to continue same basal insulin during trial participation.
6. Body Mass Index (BMI) 18.5 to 30.0 kg/m², inclusive
7. HbA1c at screening between 6.5% and 9.5% (inclusive)
8. Have clinical laboratory test results within the normal range for the population, or with abnormalities deemed clinically insignificant by the investigator.
9. Considered generally healthy (apart from type 1 diabetes and lipohypertrophy) upon completion of medical history and screening safety assessments, as judged by the Investigator
10. Have venous access sufficient to allow cannulation for blood sampling as required by the protocol

Exclusion Criteria:

1. Receipt of any medicinal product in clinical development within 60 days or 5 half-lives (if known) of the medicinal product before randomisation in this trial
2. Any history or presence of cancer, except for a history of basal cell skin cancer or squamous cell skin cancer (as judged by the Investigator)
3. Any history or presence of clinically relevant comorbidity (with the exception of conditions associated with diabetes mellitus), that may place the subject at increased risk as determined by the investigator.
4. Signs of acute illness as judged by the Investigator
5. Any serious systemic infectious disease during four weeks prior to screening, as judged by the Investigator.
6. Aspartate transaminase (AST) and/or Alanine transaminase (ALT) > 2 times the upper limit of normal
7. Estimated glomerular filtration rate (eGFR)<60 mL/min
8. Systolic blood pressure < 90 mmHg or >160 mmHg and/or diastolic blood pressure < 50 mmHg or > 95 mmHg (one repeat test will be acceptable in case of suspected white-coat hypertension)
9. Heart rate at rest outside the range of 50-90 beats per minute. This exclusion criterion also pertains to subjects being on anti-hypertensives.
10. History of severe hypoglycaemia with seizure, coma or requiring assistance of another person during the past 6 months
11. Significant history of alcoholism or drug abuse as judged by the Investigator or consuming more than 24 grams alcohol/day (for males), 12 grams alcohol/day (for females) on average
12. A positive result in the alcohol and/or urine drug screen at the screening visit
13. Tested positive for Hepatitis Bs antigen
14. Tested positive for hepatitis C antibodies. (Presence of hepatitis C antibodies will not lead to exclusion if liver function tests are normal, and a hepatitis C polymerase chain reaction is negative)
15. Positive result to the test for HIV-1/2 antibodies or HIV-1 antigen
16. Have received chronic (lasting >14 consecutive days) systemic glucocorticoid therapy (excluding topical, intra-articular, and inhaled preparations) in the past 3 months, or have received any non-topical glucocorticoid therapy within 30 days before screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Standard pharmacokinetics/pharmacodynamics (PK/PD) endpoints as applicable after injection of a rapid-acting mealtime insulin | 16 weeks
  Area under the glucose infusion rate curve (AUCGIR),0-4h: area under the glucose infusion rate curve from 0 to 4 hrs after injection of a 0.15 units/kg body weight dose of insulin lispro

SECONDARY OUTCOMES:
Effects of embrace on lipohypertrophic tissue could result in beneficial effects on volume and subsequent remodeling of the lipohypertrophic tissue histology. | From enrollment to the end of treatment of 16 weeks.
  To investigate the effect of four months of treatment with embrace® on volume (mL) of the target lipohypertrophic lesion comparing baseline to EoT in trial participants with type 1 diabetes and lipohypertrophy. To investigate the effect of four months of natural healing of a LH comparator lesion volume (mL) from baseline to EoT in trial participants with type 1 diabetes and lipohypertrophy. Measurements will be taken by ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Stoffel, Doctor, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil, Neuss, Germany

IPD SHARING:
Plan to Share IPD: No